CLINICAL TRIAL: NCT03212105
Title: A 60-seconds Personalized Mindfulness Video Exercise for Patients With Orthopedic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015P002349
Record Dates: First submitted 2017-06-06; First posted 2017-07-11 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Orthopaedic Injury; Mindfulness
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60 Second Video (Active Comparator): The mindfulness intervention is a video-flash found at http://www.pixelthoughts.co. In this exercise patients are asked to write down a concern or worry, and watch it get put into perspective within a 60 seconds time frame.
  Interventions: Behavioral: 60 Second Video
- Educational Pamphlet (Other): The educational pamphlet contains information about pain and stress, which patients will be able to read within 60 seconds.
  Interventions: Other: Educational Brochure

INTERVENTIONS:
Behavioral: 60 Second Video — The mindfulness intervention will be a video-flash found at http://www.pixelthoughts.co. In this exercise patients are asked to write down a concern or worry, and watch it get put into perspective within a 60 seconds time frame.
  Arms: 60 Second Video
Other: Educational Brochure — The educational pamphlet will contain information about pain and stress, which patients will be able to read within 60 seconds.
  Other Names: Placebo comparator
  Arms: Educational Pamphlet

SUMMARY:
The purpose of this study is to determine within a randomized controlled trial the feasibility of a 60-second acceptance based mindfulness exercise for patients with musculoskeletal pain versus usual medical care. Feasibility will be evaluated as the number of individuals approached who agree to participate and the number of individuals who drop out prior to completion of post intervention questionnaires.

The investigators aim to determine the usefulness and acceptability of the 60-second acceptance based mindfulness exercise for patients with musculoskeletal pain as compared to usual medical care. Usefulness and acceptability will be assessed with the Client Satisfaction Scale-3 (CSQ-3).

The investigators also aim to determine whether participating in a personalized 60-second acceptance based mindfulness exercise (e.g., intervention) is associated with significantly more improvement in patients' ratings of state anxiety and pain intensity (co-primary outcomes), and to determine if Distress, Anxiety, Depression and Anger (secondary outcomes) decrease compared to a brief educational pamphlet (e.g., control).

The investigators also aim to determine whether any improvements observed will maintain within a 3 month follow up.

DETAILED DESCRIPTION:
A cognitive behavioral therapy practice called Acceptance and Commitment Therapy (ACT) focuses on acceptance rather than control of thoughts, emotions and physical sensations, regardless of their quality. The crux of ACT is teaching patients to separate themselves from their thoughts (e.g., cognitive defusion) and thus decrease the importance placed on them. ACT has been successful in treating psychological disorders and emotional disturbances alone or when associated with physical illnesses, those that cause pain in particular. While ACT is effective, it may not be feasible for busy orthopedic practices. However, simple exercises that teach patients to deemphasize the importance they place on thoughts might be feasible in orthopedic settings where patients present with pain and strong emotions. An ACT exercise, delivered before the orthopedic appointment, has the potential to set the tone for a more positive experience for both patient and provider, by lowering a patient's pain intensity, state anxiety (e.g., anxiety symptoms in the present moment) as measured comprehensively by State-Trait Anxiety Inventory (STAI) questionnaire, distress, depression, anger, and anxiety, all four measured by 1 item emotional thermometers (visual scales used to rate different emotions). This exercise might help patients see ACT exercises as a helpful part of their recovery. Some might be motivated to learn more and to continue using them at home. This could improve their recovery from and adjustment to the medical condition.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Hand and Upper Extremity Service at Massachusetts General Hospital
* English fluency and literacy

Exclusion Criteria:

* Pregnant women
* Significant Axis I or II psychopathology that would interfere with participation in the study
* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Scale-3 (CSQ-3) | Day 1 after completing 60-second intervention
  The client satisfaction scale-3 (CSQ-3) is a 3 question instrument to measure satisfaction with health and human services. Responses are based on a 4-point scale. The score range is from 3-12, where higher values indicate higher satisfaction.

SECONDARY OUTCOMES:
Change in State-Trait Anxiety Inventory (STAI) | Before intervention, immediately after intervention, and 3 months after enrollment
  The STAI questionnaire measures trait and state anxiety. The questionnaire has 20 items based on a 4-point scale. A higher score is indicative of greater anxiety.
Change in Pain Intensity | Before intervention, immediately after intervention, and 3 months after enrollment
  Pain intensity as measured by ordinal rating of pain. On a scale from 0-10, where 0 is no pain and 10 is the worst pain imagined.
Change in Distress, Anxiety, Depression, and Anger | Before intervention, immediately after intervention, and 3 months after enrollment
  A visual scale using 4 emotional thermometers to measure each distress, anxiety, depression, and anger. The scale is from 0-10, where 0 means experience none of the emotion and 10 is extreme.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The video-flash mindfulness intervention — http://www.pixelthoughts.co